CLINICAL TRIAL: NCT04695067
Title: Cooperation Between NTU and NTUS: Integrated Precision Approach to Improve Baseball Skills, Tactics and Competition Performance-The Influence of Central and Peripheral Fatigue on Sports Performance and Prevention of Sports Injury
Brief Title: The Influence of Central and Peripheral Fatigue on Sports Performance and Prevention of Sports Injury
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201807126RINA
Record Dates: First submitted 2020-12-31; First posted 2021-01-05 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Central fatigue group — a fatigue protocol that pitchers need to pitch 80 trials in a simulated game

SUMMARY:
This is an observational study that assess the baseball pitchers' fatigue status. The purpose of this study is to find the pitching mechanic change and the fatigue point to provide guidance for coaches to schedule training items . It is expected that earlier detect the pitchers' fatigue point could be able to prevent overuse injury caused by compensatory actions.

DETAILED DESCRIPTION:
The expected outcomes of this study include providing more reliable scientific evidence of the effects of fatigue on baseball players' performance and movement control, which can help to improve muscle endurance and the quality of movement control. Moreover, fatigue that resulted from the prolonged practice can be reduced and recovered faster after exercise, as well as more understanding on the ideal pitching posture and compensatory action that caused by fatigue, providing a guideline for exercise training. This will not only help to prevent fatigue and reduce risk of injury, but also strengthen weak muscle groups and improve movement strategies before matches, as well as lengthen the time of being a baseball player.

ELIGIBILITY:
Inclusion Criteria:

* healthy baseball pitchers
* age between 18~35 years old

Exclusion Criteria:

* surgery history in pitching arm
* Musculoskeletal disease
* Neuromuscular disease

Ages: 18 Years to 35 Years | Sex: Male
Age Groups: Adult
Study Population: baseball pichers
Sampling Method: Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2018-10-08 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
heart rate variability (HRV) | 8 weeks
  test HRV during pitches

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Li Hsu, PhD, Principal Investigator — National Taiwan University
Locations (1):
- Taiwan, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No